CLINICAL TRIAL: NCT05392127
Title: A Single-center, Open-label, Single-arm, Fixed-sequence Study to Evaluate the Pharmacokinetic Effects of SHR0302 Tablets on Substrates of CYP3A4, CYP2C8, CYP2C9, CYP2C19 in Healthy Volunteers
Brief Title: A Pharmacokinetic Study to Evaluate the Drug Interaction Between SHR0302 and CYP Substrates in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHR0302-111
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ivarmacitinib; Midazolam; Warfarin; Vitamin K 1; repaglinide

STUDY DESIGN:
Intervention Model Description: Single-center, single arm, open-label, fixed sequence, self-control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): SHR0302 Tablets + probe drugs (Midazolam Maleate Tablets + Warfarin Sodium Tablets+ Omeprazole Enteric Capsules+ Repaglinide Tablets) + Vitamin K1 Tablets
  Interventions: Drug: SHR0302 Tablets; Drug: Midazolam Maleate Tablets; Drug: Warfarin Sodium Tablets; Drug: Omeprazole Enteric Capsules; Drug: Vitamin K1 Tablets; Drug: Repaglinide Tablets

INTERVENTIONS:
Drug: SHR0302 Tablets — SHR0302 Tablets once daily
Drug: Midazolam Maleate Tablets — Midazolam Maleate Tablets single dose
Drug: Warfarin Sodium Tablets — Warfarin Sodium Tablets single dose
Drug: Omeprazole Enteric Capsules — Omeprazole Enteric Capsules single dose
Drug: Vitamin K1 Tablets — Vitamin K1 Tablets once daily
Drug: Repaglinide Tablets — Repaglinide Tablets single dose

SUMMARY:
This is a drug-drug interaction study conducted in healthy volunteers to evaluate the pharmacokinetic effect of SHR0302 on CYP3A4, CYP2C9, CYP2C9, CYP2C19, using midazolam, s-warfarin, omeprazole, and repaglinide as probe drugs.

ELIGIBILITY:
Inclusion Criteria:

- 1.18 ≤ age ≤45, healthy male; 2.Subjects with body weight ≥ 50 kg, and 19≤BMI ≤26 kg/m2 ； 3.Subjects must agree to take effective contraceptive methods from signing informed consent to 6 months after the last administration.

Exclusion Criteria:

1. Subjects with known history or suspected of being allergic to the study drugs；
2. Participation in clinical trials of other investigational drugs or medical devices within 3 months prior to screening
3. Subjects with eGFR less than 90 mL/min/1.73m2；
4. Subjects with systolic blood pressure less than 90 mmHg or more than 140 mmHg, and/or diastolic blood pressure less than 60 mmHg or more than 90 mmHg;
5. Subjects whoes12-Lead ECG QTcF was more than 450 ms or there were other abnormalities determined by the investigator；
6. Subjects with clinically significant abnormalities in coagulation function；
7. Subjects with infectious disease；
8. Subjects with positive of urine drug screen；
9. Subjects with acute illness occurred within 4 weeks prior to the screening period;
10. Subjects who required antimicrobial therapy within 4 weeks prior to the screening period;
11. Subjects with medical history of systemic inflammatory disease, autoimmune disease, recurrent herpes zoster, disseminated herpes zoster, disseminated herpes simplex;
12. Subjects with a history of tuberculosis (TB) within six months prior to the screening period;
13. Subjects with a history of hypoglycemic episodes or fasting blood glucose less than 2.8 mmol/L during screening；
14. Subjects who took inhibitors or inducers of CYP3A4, CYP2C8, CYP2C9, or CYP2C19 within 28 days before the study;
15. Subjects with contraindications for midazolam, warfarin, omeprazole, and repaglinide.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Cmax，PK parameters of midazolam, s-warfarin, omeprazole, Repaglinide before and after oral administration of SHR0302 | Days 1-29
AUC0-t，PK parameters of midazolam, s-warfarin, omeprazole, Repaglinide before and after oral administration of SHR0302 | Days 1-29
AUC0-inf，PK parameters of midazolam, s-warfarin, omeprazole, Repaglinide before and after oral administration of SHR0302 | Days 1-29

SECONDARY OUTCOMES:
Tmax，PK parameters of midazolam, s-warfarin, omeprazole, Repaglinide before and after oral administration of SHR0302 | Days 1-29
t1/2，PK parameters of midazolam, s-warfarin, omeprazole, Repaglinide before and after oral administration of SHR0302 | Days 1-29
CL/F，PK parameters of midazolam, s-warfarin, omeprazole, Repaglinide before and after oral administration of SHR0302 | Days 1-29
Vz/F，PK parameters of midazolam, s-warfarin, omeprazole, Repaglinide before and after oral administration of SHR0302 | Days 1-29
Number of subjects with adverse events and severity of adverse events | Up to 35 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fu M, Luo L, Feng S, Lin H, Lu Z, Gu F, Fan Y, Wu B, Huang J, Shen K. Effect of SHR0302 on the pharmacokinetics of CYP3A4, CYP2C8, CYP2C9 and CYP2C19 probe substrates in healthy volunteers: A cocktail analysis. Br J Clin Pharmacol. 2023 Dec;89(12):3659-3668. doi: 10.1111/bcp.15856. Epub 2023 Aug 22. PMID 37464978